CLINICAL TRIAL: NCT02547935
Title: An Exploratory Phase II/III, Randomized, Double-blind, Placebo Controlled, Parallel Design Study to Evaluate the Efficacy, Safety and Pharmacodynamics of Dapagliflozin and Dapagliflozin in Combination With Saxagliptin in CKD Patients With Type 2 Diabetes Mellitus and Albuminuria Treated With ACEi or ARB
Brief Title: A Study to Evaluate the Effect of Dapagliflozin With and Without Saxagliptin on Albuminuria, and to Investigate the Effect of Dapagliflozin and Saxagliptin on HbA1c in Patients With Type 2 Diabetes and CKD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1690C00023
Record Dates: First submitted 2015-08-31; First posted 2015-09-14 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes Mellitus, CKD and Albuminuria
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Albuminuria | interventions — dapagliflozin; saxagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dapagliflozin 10mg (Experimental): Tablets administered orally once daily for 24 weeks
  Interventions: Drug: Dapagliflozin 10 mg
- Dapagliflozin 10mg + Saxagliptin 2.5mg (Experimental): Tablets administered orally once daily for 24 weeks
  Interventions: Drug: Saxagliptin 2.5 mg
- Placebo (Placebo Comparator): Tablets administered orally once daily for 24 weeks
  Interventions: Drug: Matching Placebo for Dapagliflozin 10 mg and Saxagliptin 2.5mg

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — Tablets administered orally once daily for 24 weeks.
  Other Names: Forxiga™
  Arms: Dapagliflozin 10mg
Drug: Saxagliptin 2.5 mg — Tablets administered orally once daily for 24 weeks.
  Other Names: Onglyza™
  Arms: Dapagliflozin 10mg + Saxagliptin 2.5mg
Drug: Matching Placebo for Dapagliflozin 10 mg and Saxagliptin 2.5mg — Tablets administered orally once daily for 24 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this clinical research study is to determine whether dapagliflozin alone or in combination with saxagliptin can decrease albuminuria and improve glycemic control in patients with Type 2 diabetes, albuminuria and renal impairment (CKD). The study is planned to randomize a total of 450 patients (150 patients per treatment arm)

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Female or male aged ≥18 years
* History of type 2 diabetes mellitus for more than 12 months
* HbA1c≥7.0% and ≤11.0%
* Stable antidiabetic treatment during the last 12 weeks up to randomization
* eGFR 25-75 mL/minute/1.73m2, inclusive
* Micro or macroalbuminuria (UACR 30 - 3500 mg/g)
* Treatment with ACE inhibitor or an ARB for at least 3 months prior to screening
* Body mass index between 20 and 45 kg/m2

Exclusion Criteria:

* Any of the following CV/Vascular Diseases within 3 month prior to signing the consent at Visit 1:

  * Myocardial infarction
  * cardiac surgery or revascularization (CABG/PTCA)
  * unstable angina
  * unstable HF
  * New York Heart Association (NYHA) Class III-IV
  * transient ischemic attack (TIA) or significant cerebrovascular disease
  * unstable or previously undiagnosed arrhythmia
* Significant hepatic disease, including, but not limited to, chronic active hepatitis and/or severe hepatic insufficiency
* Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) > 3X ULN
* Total Bilirubin (TB) >2 mg/dL (34.2 μmol/L)
* History of acute kidney injury requiring renal replacement therapy (dialysis or ultrafiltration) or any biopsy or imaging verifying intercurrent kidney disease other than diabetic nephropathy or diabetic nephropathy with nephrosclerosis
* Ongoing treatment with a SGLT2 inhibitor, GLP-1 agonist or DPP4 inhibitors
* Any condition which, in the judgment of the Investigator, may render the patient unable to complete the study or which may pose a significant risk to the patient or patient suspected or with confirmed poor protocol or medication compliance

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (98):
- United States (37):
  - Research Site, Peoria, Arizona
  - Research Site, Chula Vista, California
  - Research Site, Concord, California
  - Research Site, El Centro, California
  - Research Site, La Mesa, California
  - Research Site, Long Beach, California
  - Research Site, Los Gatos, California
  - Research Site, North Hollywood, California
  - Research Site, Riverside, California
  - Research Site, San Diego, California
  - Research Site, San Dimas, California
  - Research Site, Hollywood, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Bangor, Maine
  - Research Site, Kansas City, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Springfield Gardens, New York
  - Research Site, The Bronx, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Brownsville, Texas
  - Research Site, Cypress, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Burke, Virginia
  - Research Site, Richmond, Virginia
- Australia (4):
  - Research Site, Box Hill
  - Research Site, Campbelltown
  - Research Site, Geelong
  - Research Site, Herston
- Canada (10):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, Ajax, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Jérôme, Quebec
  - Research Site, Sherbrooke, Quebec
- Japan (12):
  - Research Site, Chūōku
  - Research Site, Hachioji-shi
  - Research Site, Higashiosaka-shi
  - Research Site, Kisarazu-shi
  - Research Site, Kyoto
  - Research Site, Neyagawa
  - Research Site, Nishinomiya-shi
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Toyonaka-shi
- Mexico (7):
  - Research Site, Aguascalientes
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Querétaro
  - Research Site, Zapopan
  - Research Site, Zapopan, Jalisco
- South Africa (8):
  - Research Site, Benoni
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Kuilsrivier
  - Research Site, Mamelodi East
  - Research Site, Muckleneuk
  - Research Site, Paarl
  - Research Site, Pretoria
- South Korea (8):
  - Research Site, Ansan-si
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Daejeon
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Wŏnju
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Sabadell (Barcelona)
  - Research Site, Santiago(A Coruña)
  - Research Site, Valencia
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung Hsien
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Yongkang District

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Koshino A, Neuen BL, Jongs N, Pollock C, Greasley PJ, Andersson EM, Hammarstedt A, Karlsson C, Langkilde AM, Wada T, Heerspink HJL. Effects of dapagliflozin and dapagliflozin-saxagliptin on erythropoiesis, iron and inflammation markers in patients with type 2 diabetes and chronic kidney disease: data from the DELIGHT trial. Cardiovasc Diabetol. 2023 Nov 28;22(1):330. doi: 10.1186/s12933-023-02027-8. PMID 38017482
- [Derived] Pollock C, Stefansson B, Reyner D, Rossing P, Sjostrom CD, Wheeler DC, Langkilde AM, Heerspink HJL. Albuminuria-lowering effect of dapagliflozin alone and in combination with saxagliptin and effect of dapagliflozin and saxagliptin on glycaemic control in patients with type 2 diabetes and chronic kidney disease (DELIGHT): a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2019 Jun;7(6):429-441. doi: 10.1016/S2213-8587(19)30086-5. Epub 2019 Apr 13. PMID 30992195
- See also: D1690c00023_CSP_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3763&filename=D1690c00023_CSP_Redacted.pdf
- See also: D1690c00023_SAP_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3763&filename=D1690c00023_SAP_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Chronic Kidney Disease and Type 2 Diabetes Mellitus with micro- or macro-albuminuria and treated with ACEi or ARB were enrolled into an international, multi-centre study from 21 Sep 2015. The last patient's last visit was 18 May 2018.
Pre-assignment Details: Enrolled patients were screened during a 4-week single-blind placebo lead-in period. Patients who met all of the inclusion and none of the exclusion criteria in this period were eligible to be randomised into the 24-week double-blind placebo-controlled treatment period.
Groups:
- Dapagliflozin 10 mg + Saxagliptin 2.5 mg: Dapagliflozin 10 milligram (mg) and saxagliptin 2.5 mg tablets were taken orally, once daily (in the morning) for 24 weeks.
- Dapagliflozin 10 mg: Dapagliflozin 10 mg tablets were taken orally, once daily (in the morning) for 24 weeks. Patients also took placebo tablets to match saxagliptin.
- Placebo: Placebo tablets to match both active products (dapagliflozin and saxagliptin) were taken orally, once daily (in the morning) for 24 weeks.
Period: Overall Study
Arm/Group | Dapagliflozin 10 mg + Saxagliptin 2.5 mg | Dapagliflozin 10 mg | Placebo
Started (Patients randomised to 24-week double-blind treatment period.) | 155 | 145 | 148
Received Treatment | 152 | 145 | 148
Full Analysis Set | 152 | 144 | 148
Safety Analysis Set | 152 | 145 | 148
Completed | 150 | 137 | 143
Not Completed | 5 | 8 | 5
Not completed — Other | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 4
Not completed — Screen Failure | 2 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Death | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for all randomised patients.
Groups:
- Dapagliflozin 10 mg + Saxagliptin 2.5 mg: Dapagliflozin 10 mg and saxagliptin 2.5 mg tablets were taken orally, once daily (in the morning) for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 10 mg + Saxagliptin 2.5 mg | Dapagliflozin 10 mg | Placebo | Total
Number analyzed (Participants) | 155 | 145 | 148 | 448
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.21) | 64.7 (8.61) | 64.7 (8.53) | 64.4 (8.78)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 78 | 64 | 68 | 210
  >=65 years | 77 | 81 | 80 | 238
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 43 | 43 | 131
  Male | 110 | 102 | 105 | 317
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 32 | 38 | 112
  Not Hispanic or Latino | 113 | 113 | 110 | 336
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 77 | 55 | 64 | 196
  Black or African American | 8 | 7 | 11 | 26
  Asian | 57 | 67 | 53 | 177
  Native Hawaiian or other Pacific Islander | 1 | 2 | 1 | 4
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Other | 12 | 13 | 18 | 43

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Glycosylated Haemoglobin (HbA1c): Comparison of Dapagliflozin 10 mg Plus Saxagliptin 2.5 mg and Placebo at Week 24
Description: HbA1c was analysed at baseline and every 4 weeks during the 24-week treatment period. Only measurements prior to rescue or treatment discontinuation were analysed. The adjusted mean change from baseline at Week 24 was analysed using a mixed model repeated measures (MMRM) model.
Time Frame: Baseline and Week 24
Population: Patients from the Full Analysis Set (all randomised patients who took at least 1 dose of double-blind study drug and had a non missing baseline value and at least one post-baseline efficacy variable value) with non-missing baseline and Week 24 values for HbA1c.
Measure: Least Squares Mean (Standard Error); unit: Percentage of Glycoslyated HbA1c
Arm/Group | Dapagliflozin 10 mg + Saxagliptin 2.5 mg | Placebo
Number analyzed (Participants) | 151 | 145
Percentage of Glycoslyated HbA1c | -0.85 (0.09) | -0.27 (0.09)
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg + Saxagliptin 2.5 mg vs Placebo; A longitudinal repeated measures analysis included the fixed categorical effects of treatment, week, randomisation stratification factor (i.e. anti-diabetic treatment strata), and treatment-by-week interaction, as well as the continuous fixed covariates of baseline measurement and baseline measurement-by-week interaction; Test type: Superiority; p < 0.001, MMRM — Statistical significance level = 0.025; Difference in adjusted mean change = -0.58, 95% CI 2-sided [-0.80 to -0.37], Standard Error of Mean 0.11

2. Primary Outcome: Adjusted Mean Percent Change From Baseline in Urine Albumin-to-Creatinine Ratio (UACR) at Week 24
Description: UACR was analysed at baseline and every 4 weeks during the 24-week treatment period. All measurements regardless of rescue medication or treatment discontinuation were analysed. UACR values were first transformed to logarithms and the results were based on exponentiation of model estimates and expressed as adjusted mean percent change from baseline at Week 24.
Time Frame: Baseline and Week 24
Population: Patients from the Full Analysis Set with non-missing baseline and Week 24 values for UACR.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Dapagliflozin 10 mg + Saxagliptin 2.5 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 151 | 140 | 144
Percent change | -39.1 (5.1) | -22.4 (6.6) | -1.8 (8.3)
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg + Saxagliptin 2.5 mg vs Placebo; A longitudinal repeated measures model of the logarithms of the post-baseline to baseline ratios included the fixed categorical effects of treatment, week, treatment-by-week interaction, and randomisation stratification factor (i.e. anti-diabetic treatment strata), as well as the continuous fixed covariates of log-baseline UACR value and log-baseline UACR value-by-week interaction; Test type: Superiority; p < 0.001, MMRM — Statistical significance level = 0.025; Difference in adjusted mean change = -38.0, 95% CI 2-sided [-48.2 to -25.8], Standard Error of Mean 5.7
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.011, MMRM — Statistical significance level = 0.025; Difference in adjusted mean change = -21.0, 95% CI 2-sided [-34.1 to -5.2], Standard Error of Mean 7.3

3. Secondary Outcome: Adjusted Mean Percent Change From Baseline in Total Body Weight at Week 24
Description: Total body weight was measured in kilograms (kg) at baseline and at Week 1 then every 4 weeks during the 24-week treatment period. All measurements regardless of rescue medication or treatment discontinuation were analysed. Total body weight values were first transformed to logarithms and the results were based on exponentiation of model estimates and expressed as adjusted mean percent change from baseline at Week 24.
Time Frame: Baseline and Week 24
Population: Patients from the Full Analysis Set with non-missing baseline and Week 24 values for total body weight.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Dapagliflozin 10 mg + Saxagliptin 2.5 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 152 | 144 | 148
Percent change | -0.65 (0.55) | -1.48 (0.56) | -0.61 (0.56)
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg + Saxagliptin 2.5 mg vs Placebo; A longitudinal repeated measures model of the logarithms of the post-baseline to baseline ratios included the fixed categorical effects of treatment, week, treatment-by-week interaction, and randomisation stratification factor (i.e. anti-diabetic treatment strata), as well as the continuous fixed covariates of log-baseline total body weight value and log-baseline total body weight value-by-week interaction; Test type: Superiority; p = 0.953, MMRM — Statistical significance level = 0.025; Difference in adjusted mean change = -0.04, 95% CI 2-sided [-1.32 to 1.26], Standard Error of Mean 0.66
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.193, MMRM — Statistical significance level = 0.025; Difference in adjusted mean change = -0.87, 95% CI 2-sided [-2.17 to 0.44], Standard Error of Mean 0.66

4. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: FPG was analysed at baseline and Week 1 then every 4 weeks during the 24-week treatment period. Only measurements prior to rescue or treatment discontinuation were analysed. The adjusted mean change from baseline at Week 24 was analysed using a MMRM model.
Time Frame: Baseline and Week 24
Population: Patients from the Full Analysis Set with non-missing baseline and Week 24 values for FPG.
Measure: Least Squares Mean (Standard Error); unit: mg/decilitre (dL)
Arm/Group | Dapagliflozin 10 mg + Saxagliptin 2.5 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 152 | 144 | 147
mg/decilitre (dL) | -17.2 (5.2) | -13.1 (5.4) | -11.2 (5.5)
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg + Saxagliptin 2.5 mg vs Placebo; A longitudinal repeated measures analysis included the fixed categorical effects of treatment, week, randomisation stratification factor (i.e.anti-diabetic treatment strata), and treatment-by-week interaction, as well as the continuous fixed covariates of baseline measurement and baseline measurement-by-week interaction; Test type: Superiority; p = 0.298, MMRM — Statistical significance level = 0.025; Difference in adjusted mean change = -6.1, 95% CI 2-sided [-17.5 to 5.4], Standard Error of Mean 5.8
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.746, MMRM — Statistical significance level = 0.025; Difference in adjusted mean change = -1.9, 95% CI 2-sided [-13.6 to 9.8], Standard Error of Mean 5.9

5. Secondary Outcome: Percentage of Patients Achieving at Least 30% Reduction in UACR at Week 24
Description: The percentage of patients meeting the criteria of at least a 30% reduction in UACR, was analysed using a logistic regression model. If no measurement was available at Week 24 the last available post-baseline measurement was carried forward (Last Observation Carried Forward [LOCF]).
Time Frame: From baseline up to Week 24
Population: Patients from the Full Analysis Set with non-missing baseline and at least one post-baseline UACR value.
Measure: Number; unit: Percentage of patients
Arm/Group | Dapagliflozin 10 mg + Saxagliptin 2.5 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 152 | 144 | 148
Percentage of patients | 57.0 | 45.0 | 31.3
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg + Saxagliptin 2.5 mg vs Placebo; Logistic regression model analysis with adjustment for baseline UACR and pooled randomisation strata; Test type: Superiority; p < 0.001, Regression, Logistic — Statistical significance level = 0.025; Odds Ratio (OR) = 2.98, 95% CI 2-sided [1.8 to 4.8]
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Placebo; Logistic regression model analysis with adjustment for baseline UACR and pooled randomisation strata; Test type: Superiority; p = 0.013, Regression, Logistic — Statistical significance level = 0.025; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.1 to 3.0]

6. Secondary Outcome: Percentage of Patients Achieving a Reduction in HbA1c of Less Than 7.0% at Week 24
Description: The percentage of patients meeting the criteria of a less than 7% reduction in HbA1c, was analysed using a logistic regression model. If no measurement was available at Week 24 the last available post-baseline measurement was carried forward (LOCF). Only measurements prior to rescue or treatment discontinuation were analysed.
Time Frame: From baseline to Week 24
Population: Patients from the Full Analysis Set with non-missing baseline and at least one post-baseline HbA1c value.
Measure: Number; unit: Percentage of patients
Arm/Group | Dapagliflozin 10 mg + Saxagliptin 2.5 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 152 | 144 | 148
Percentage of patients | 35.1 | 15.0 | 10.3
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg + Saxagliptin 2.5 mg vs Placebo; Logistic regression model analysis with adjustment for baseline HbA1c and pooled randomisation strata; Test type: Superiority; p < 0.001, Regression, Logistic — Statistical significance level = 0.025; Odds Ratio (OR) = 5.43, 95% CI 2-sided [2.6 to 11.2]
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Placebo; Logistic regression model analysis with adjustment for baseline HbA1c and pooled randomisation strata; Test type: Superiority; p = 0.167, Regression, Logistic — Statistical significance level = 0.025; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.8 to 3.8]

7. Secondary Outcome: Adjusted Mean Change From Baseline in Seated Systolic Blood Pressure (SBP) at Week 24
Description: Seated SBP was analysed at baseline, Week 1 and every 4 weeks during the 24-week treatment period. All measurements regardless of rescue medication or treatment discontinuation were analysed. The adjusted mean change from baseline at Week 24 was analysed using a MMRM model.
Time Frame: Baseline and Week 24
Population: Patients from the Full Analysis Set with non-missing baseline and Week 24 values for SBP.
Measure: Least Squares Mean (Standard Error); unit: Millimetre of mercury (mmHg)
Arm/Group | Dapagliflozin 10 mg + Saxagliptin 2.5 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 152 | 144 | 147
Millimetre of mercury (mmHg) | -8.8 (1.6) | -6.9 (1.7) | -4.1 (1.7)
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg + Saxagliptin 2.5 mg vs Placebo; A longitudinal repeated measures model of the logarithms of the post-baseline to baseline ratios, included the fixed categorical effects of treatment, week, treatment-by-week interaction, and randomisation strata, as well as the continuous fixed covariates of log-baseline SBP value and log-baseline SBP value-by-week interaction; Test type: Superiority; p = 0.009, MMRM — Statistical significance level = 0.025; Difference in adjusted mean change = -4.8, 95% CI 2-sided [-8.3 to -1.2], Standard Error of Mean 1.8
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.122, MMRM — Statistical significance level = 0.025; Difference in adjusted mean change = -2.8, 95% CI 2-sided [-6.4 to 0.8], Standard Error of Mean 1.8

8. Secondary Outcome: Adjusted Mean Change From Baseline in HbA1c: Comparison of Dapagliflozin 10 mg and Placebo at Week 24
Description: HbA1c was analysed at baseline and every 4 weeks during the 24-week treatment period. Only measurements prior to rescue or treatment discontinuation were analysed. The adjusted mean change from baseline at Week 24 was analysed using a MMRM model.
Time Frame: Baseline and Week 24
Population: Patients from the Full Analysis Set with non-missing baseline and Week 24 values for HbA1c.
Measure: Least Squares Mean (Standard Error); unit: Percentage of Glycoslyated HbA1c
Arm/Group | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 140 | 145
Percentage of Glycoslyated HbA1c | -0.43 (0.09) | -0.27 (0.09)
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.142, MMRM — Statistical significance level = 0.025; Difference in adjusted mean change = -0.16, 95% CI 2-sided [-0.38 to 0.05], Standard Error of Mean 0.11

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are reported from Day 1 of the 24-week double-blind treatment period. Non-serious AEs were included up to the last day of double-blind treatment + 4 days. Serious AEs were included up to the last day of double-blind treatment + 30 days, giving a total maximum time frame of 28 weeks.
Description: The Safety Analysis Set consisted of all patients who received at least 1 dose of study drug during the 24-week double-blind treatment period.
Groups:
- Placebo: Placebo tablets to match both active products (dapagliflozin and saxagliptin)were taken orally, once daily (in the morning) for 24 weeks.
Arm/Group | Dapagliflozin 10 mg + Saxagliptin 2.5 mg | Dapagliflozin 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/152 | 1/145 | 0/148
Serious Adverse Events (participants affected / at risk) | 12/152 | 12/145 | 16/148
Other Adverse Events (participants affected / at risk) | 12/152 | 18/145 | 8/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 10 mg + Saxagliptin 2.5 mg (N=152) | Dapagliflozin 10 mg (N=145) | Placebo (N=148)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Emphysematous pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Genital infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 10 mg + Saxagliptin 2.5 mg (N=152) | Dapagliflozin 10 mg (N=145) | Placebo (N=148)
Influenza (Infections and infestations) | 2 (2) | 8 (8) | 2 (2)
Nasopharyngitis (Infections and infestations) | 10 (12) | 10 (11) | 6 (6)

LIMITATIONS AND CAVEATS:
Anomalous data at 1 site was identified following completion of the study. All data from this site were excluded from the full analysis following an audit; the findings led the sponsor to believe the site did not comply with the principles of GCP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT02547935/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT02547935/SAP_001.pdf